CLINICAL TRIAL: NCT05156970
Title: A Multicenter, Prospective, Double-Cohort Phase II Clinical Study of Camrelizumab in Combination With Docetaxel and Platinum or Apatinib Mesylate as First-Line Treatment for Recurrent or Metastatic Head and Neck Squamous Cell Carcinoma
Brief Title: Camrelizumab in Combination With Chemotherapy or Apatinib Mesylate as First-Line Treatment for R/M HNSCC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University (Other)
Responsible Party: Principal Investigator, ren guoxin, Dr., Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MA-HNC-II-002
Record Dates: First submitted 2021-06-21; First posted 2021-12-14 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Recurrent Head and Neck Squamous Cell Carcinoma; Metastatic Head and Neck Squamous Cell Carcinoma
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — camrelizumab; Cisplatin; Docetaxel; apatinib; Carboplatin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Camrelizumab + Chemotherapy (Experimental): Participants receive Camrelizumab 200 mg intravenously (IV) on Day 1 of each 3-week cycle for up to 24 months;plus cisplatin 75 mg/m^2 IV or carboplatin at a target area under the curve of 5 (AUC 5) IV, per Investigator's choice, on Day 1 of each 3-week cycle (6 cycle maximum); plus docetaxel 75 mg/m^2 IV on Day 1 of each 3-week cycle (6 cycle maximum).
  Interventions: Drug: Camrelizumab; Drug: Cisplatin; Drug: Docetaxel; Drug: Carboplatin
- Camrelizumab +Apatinib mesylate (Experimental): Participants receive Camrelizumab 200 mg intravenously (IV) on Day 1 of each 3-week cycle for up to 24 months;plus Apatinib 250mg qd for up to 24 months.
  Interventions: Drug: Camrelizumab; Drug: Apatinib Mesylate

INTERVENTIONS:
Drug: Camrelizumab — Camrelizumab 200 mg IV on Day 1 of each 3-week cycle for up to 24 months
  Other Names: AiRuiKa™; SHR-1210
Drug: Cisplatin — Cisplatin 75 mg/m^2 or Carboplatin AUC5 IV on Day 1 of each 3-week cycle (4 to 6 cycle maximum)
  Other Names: Platinol
  Arms: Camrelizumab + Chemotherapy
Drug: Docetaxel — Docetaxel 75 mg/m^2 IV on Day 1 of each 3-week cycle (4 to 6 cycle maximum)
  Other Names: DTX
  Arms: Camrelizumab + Chemotherapy
Drug: Apatinib Mesylate — Apatinib 250mg qd for up to 24 months
  Other Names: YN968D1
  Arms: Camrelizumab +Apatinib mesylate
Drug: Carboplatin — Carboplatin at a target AUC 5 IV on Day 1 of each 3-week cycle (6 cycle maximum)
  Other Names: Paraplatin
  Arms: Camrelizumab + Chemotherapy

SUMMARY:
This study is the first clinical study of first-line treatment of head and neck squamous cell carcinoma with drugs targeting VEGF signaling pathway combined with PD-1 inhibitors in China, which explores the new combination therapies urgently needed in clinical practice and lays a foundation for subsequent studies, with important scientific research significance and clinical value.

DETAILED DESCRIPTION:
Head and neck cancer is the sixth most common cancer in the world, with more than 550,000 cases and 300,000 deaths worldwide each year. About 75,000 Chinese suffer from head and neck cancer each year, and currently, there are a total of 176,000 patients with head and neck cancer in China. More than 95% of head and neck cancers are squamous cell carcinomas, and head and neck squamous cell carcinoma (SCCHN) disrupts and affects the patient's appearance and basic physiological functions, sensory functions, and language functions, thus affecting the patient's quality of life. Most head and neck squamous cell carcinomas are incurable, and they will develop local recurrence and metastasis.

More than 60% of patients with head and neck squamous cell carcinoma have stage III or IV disease characterized by large size tumors with marked local invasion, evidence of metastasis to regional lymph nodes, or both. Locally advanced head and neck cancer has a high risk of local recurrence and distant metastasis and a poor prognosis. Over the past 20 years, multimodal treatment approaches have steadily improved cure rates while striving to maintain patient function and quality of life.

Currently, there are a large number of ongoing clinical trials that combine targeted therapies and immunotherapies. The basic rationale behind these combinations is that they combine different immunological and tumor biological mechanisms to enhance antitumor activity; in addition, some evidence suggests that targeted therapies can enhance certain aspects of the "cancer-immune cycle" (e.g., tumor antigenicity, T cell priming/trafficking/infiltration, etc.) to synergistically enhance immunotherapy.

This clinical study involved Recombinant Humanized Anti-PD-1 Monoclonal Antibody Injection (Camrelizumab), a Class 1 new therapeutic biological product developed by Jiangsu Hengrui Medicine Co., Ltd., which was approved by NMPA in May 2019 for the treatment of relapsed or refractory classical Hodgkin's lymphoma, by NMPA in March 2020 for the treatment of patients with advanced hepatocellular carcinoma who have received sorafenib and/or oxaliplatin-based systemic chemotherapy, and in June 2020 for the second-line treatment of esophageal squamous cell carcinoma and first-line treatment of non-squamous non-small cell lung cancer.

Preclinical study data showed that camrelizumab had comparable in vivo efficacy and safety compared with similar drugs abroad. Since 2015, Hengrui has simultaneously carried out a number of phase I/II clinical trials in Australia and China to preliminarily verify the safety, tolerability and efficacy of camreibizumab in the treatment of advanced solid tumors.

This clinical study also involved apatinib mesylate developed by Jiangsu Hengrui Medicine Co., Ltd. and marketed in 2014. Apatinib mesylate is a small molecule targeted drug, a vascular endothelial growth factor receptor (VEGFR) tyrosine kinase inhibitor, which exerts anti-angiogenic effect mainly by inhibiting VEGFR to treat malignant tumors. Preclinical studies have shown that its anti-tumor effect is superior to that of similar drugs. In 2014, apatinib mesylate has been used in patients with advanced gastric or gastro-esophageal junction adenocarcinoma who have progressed or relapsed after at least 2 prior systemic chemotherapies.

ELIGIBILITY:
Inclusion Criteria:

1. Newly diagnosed recurrent or metastatic head and neck squamous cell carcinoma which is histologically or cytologically confirmed, and unable to be cured by local treatment (the primary site of the tumor is the oropharynx, oral cavity, hypopharynx and larynx), recurrence or metastasis stage did not receive any anti-tumor systemic therapy (allowed as part of the treatment of locally advanced tumors, and it has been more than 6 months from the end of treatment to signing the informed consent);
2. ECOG score of 0 or 1;
3. At least one measurable lesion according to RECIST1.1 criteria.
4. Tumor tissue with PD-L1 detection (paraffin specimens or fresh tumor tissue within 2 years) can be provided; Patients with Oropharyngeal cancer should provide P16 detection status by using IHC method;
5. Patients with a history of brain/meningeal metastasis must be treated with local therapy (surgery/radiotherapy) before the start of the study, and clinically stable for at least 3 months (corticosteroids are allowed before the first dose of the study drug, but need to be discontinued 2 weeks before the start of the study drug); The subjects voluntarily joined the study, signed the informed consent form, had good compliance, and cooperated with the follow-up.

Exclusion Criteria:

1. Progression within 6 months after systemic treatment for locally advanced head and neck squamous cell carcinoma;
2. Previous history of primary tumor of nasopharyngeal carcinoma;
3. Intolerable to platinum-based therapy;
4. Previous treatment with platinum-based regimen and disease progression;
5. Patients who participated in or were participating in other drug/therapy clinical trials 4 weeks before the first dose of study drug;
6. Patients who underwent major surgery or had not recovered from the side effects of this surgery; Patients who has accepted live vaccination, immunotherapy, or patients who underwent radiotherapy within 2 weeks;
7. Patients who received any other anti-tumor treatment;
8. Patients who are using immunosuppressive agents, or systemic hormone therapy to achieve the purpose of immunosuppression (dose > 10 mg/day prednisone or other effective hormones), and continue to use 2 times before enrollment;
9. History of other malignant tumors within the past 5 years, except cured cutaneous basal cell carcinoma, cutaneous squamous cell carcinoma, early prostate cancer and cervical carcinoma in situ;
10. Patients who have received hematopoietic stimulating factors, such as granulocyte colony-stimulating factor (G-CSF), erythropoietin and other treatments before the first dose of study drug;
11. Prior treatment with PD-1/PD-L1/PD-L2/CTLA-4 antibodies or activating or inhibiting drugs against T cell receptors (e.g., OX40, CD137);
12. Presence of active or uncontrolled metastatic central nervous system tumor lesions diagnosed by imaging;
13. Positive test results for HIV antibody or Treponema pallidum antibody;
14. Known to be allergic to recombinant humanized PD-1 monoclonal antibody drugs and their components;
15. Active pulmonary disease (interstitial pneumonia, pneumonia, obstructive pulmonary disease, asthma) or history of active pulmonary tuberculosis;
16. Patients who have received re-radiotherapy in the head and neck position (including cervical, supraclavicular and subclavian lymph nodes) within 6 months before enrollment;
17. Patients who have tumor encasement, invasion or infiltration of large blood vessels, invasion of the skin or mucosal cavity, or ulceration and bleeding of tumor lesions;
18. Patients who have previously received VEGF/VEGFR-targeted anti-vascular drug therapy;
19. Patients who are known to be allergic to Apatinib mesylate and any excipients of it;
20. Patients who are suffering from hypertension, and cannot be well controlled by antihypertensive drug therapy (systolic blood pressure ≥ 140 mmHg or diastolic blood pressure ≥ 90 mmHg);
21. Patients who have any condition affecting the swallowing of drugs by subjects, and any condition affecting the disposition process (absorption, distribution, metabolism or excretion) of the test drug in the body;
22. Patients who have coagulation abnormalities (INR > 2.0, PT > 16 s), with bleeding tendency or receiving thrombolytic or anticoagulant therapy. Prophylactic use of low-dose aspirin, low-molecular-weight heparin is permitted.
23. Patients who had clinically significant bleeding symptoms or clear bleeding tendency within 3 months before enrollment, such as pertussis/hemoptysis of 2.5ml or more, gastrointestinal bleeding, esophageal and gastric varices at risk of bleeding, hemorrhagic gastric ulcer or suffering from vasculitis, etc.
24. Known inherited or acquired bleeding or thrombotic tendencies (e.g., hemophilia, coagulopathy, thrombocytopenia, etc.)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2021-06-24 (Actual); Primary Completion 2024-06-24 (Actual); Study Completion 2025-06-24 (Actual)

PRIMARY OUTCOMES:
Overall Survival (OS) in All Participants | 12 months
  OS was defined as the time from randomization to death due to any cause. Participants without documented death at the time of the final analysis were censored at the date of the last follow-up.

SECONDARY OUTCOMES:
Progression Free Survival Per RECIST 1.1 | 12 months
  PFS was defined as the time from randomization to the first documented PD per RECIST 1.1, or death due to any cause, whichever occurred first. Per RECIST 1.1, PD was defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum had to demonstrate an absolute increase of ≥5 mm. The appearance of one or more new lesions was also considered PD.
Objective Response Rate Per RECIST 1.1 | 12 months
  ORR was defined as the percentage of participants in the analysis population who have a Complete Response (CR: disappearance of all target lesions) or a Partial Response (PR: ≥30% decrease in the sum of diameters of target lesions) per RECIST 1.1.
Duration of Response Per RECIST 1.1 | 24 months
  Duration of response-defined as the time from first documented complete or partial response to radiographically confirmed disease progression or death from any cause, whichever occurred first.
ORR in Participants With PD-L1 CPS ≥1 | 12 months
  ORR was defined as the percentage of participants in the analysis population who have a Complete Response (CR: disappearance of all target lesions) or a Partial Response (PR: ≥30% decrease in the sum of diameters of target lesions) per RECIST 1.1.
ORR in Participants With PD-L1 CPS ≥20 | 12 months
  ORR was defined as the percentage of participants in the analysis population who have a Complete Response (CR: disappearance of all target lesions) or a Partial Response (PR: ≥30% decrease in the sum of diameters of target lesions) per RECIST 1.1.
DOR in Participants With PD-L1 CPS ≥1 | 24 months
  Duration of response-defined as the time from first documented complete or partial response to radiographically confirmed disease progression or death from any cause, whichever occurred first.
DOR in Participants With PD-L1 CPS ≥20 | 12 months
  Duration of response-defined as the time from first documented complete or partial response to radiographically confirmed disease progression or death from any cause, whichever occurred first.
Number of Participants Experiencing an Adverse Event (AE). | 12 months
  An AE was defined as any untoward medical occurrence in a participant administered a pharmaceutical product and which did not necessarily have to have a causal relationship with this treatment. An AE could therefore be any unfavourable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product or protocol-specified procedure, whether or not considered related to the medicinal product or protocol-specified procedure. Any worsening of a pre-existing condition that was temporally associated with the use of the Sponsor's product was also an AE. The number of participants that experienced at least one AE was reported for each treatment arm.
Quality of life（EORTC QLQ-C30 scale） | 12 months
  The EORTC-QLQ-C30 is a 30-item questionnaire developed to assess the quality of life of cancer patients. Participant responses to the GHS question "How would you rate your overall health during the past week?" (Item 29) and the QoL question "How would you rate your overall quality of life during the past week?" (Item 30) were scored on a 7-point scale (1=Very Poor to 7=Excellent).

CONTACTS AND LOCATIONS:
Overall Officials: Chenping Zhang, M.D., Principal Investigator — the Ninth People's Hospital Affiliated to Shanghai Jiao Tong University School of Medicine
Locations (1):
- the Ninth People's Hospital Affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai, China

IPD SHARING:
Plan to Share IPD: No